CLINICAL TRIAL: NCT04301700
Title: Effects of Progressive Muscle Relaxation and Mindfulness Meditation on Dyspnea, Fatigue and Care Dependency in Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Study
Brief Title: Effects of Progressive Muscle Relaxation and Mindfulness Meditation in Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aylin Helvaci, Research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2408
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: COPD; Mediation; Fatigue; Symptoms and Signs
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Negotiating; Fatigue; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- relaxation (Experimental): The progressive muscle relaxation intervention, designed by Jacobson (1987), will be consist of sessions involving straining and relaxing all muscle groups from head to foot with deep breathing and last for 20 min. The patients will be asked to tense a very muscle group for 5 s and relax after counting up to 10 s while breathing out. In this way, facial, head, neck, shoulders, arms, chest, abdomen, legs, hips, feet and fingers muscles are stretched and relaxed on purpose for relaxing in patients with COPD.
  Interventions: Behavioral: mindfullness and relaxation
- mindfulness meditation (Experimental): The research team closely will be following the mindfulness meditation intervention, developed by Kabat-Zinn, Lipworth, and Burney (1985), which is a part of the mindfulness-based stress reduction program. Mindfulness meditation is including interventions such as yoga, body scan, walking meditation, and sitting meditations. In the present study, the researchers will prefer sitting meditation. In this context, the second co-author will want patients to sit up in the chair in an upright and comfortable position. The patients will focus on deep breathing and felled the breath flowing throughout their body during the interventions that will last for 20 min in each session.
  Interventions: Behavioral: mindfullness and relaxation
- Control (No Intervention): Patients will continue to receive standard nursing care and no further intervention will be made during the research.

INTERVENTIONS:
Behavioral: mindfullness and relaxation — three arms: mindfullness and relaxation
  Arms: mindfulness meditation; relaxation

SUMMARY:
Patients with COPD will be entered. Participants will be randomized to one of three study arms: Arm 1: meditation; Arm 2: relaxation; Arm 3: Control. Hypothesis: Progressive muscle relaxation and mindfulness meditation will decrease severity of dyspnea, fatigue and care dependency.

DETAILED DESCRIPTION:
Previous reports have revealed that progressive muscle relaxation and meditation are decreasing symptoms burden in chronic disease. On the other hand, no study has been conducted to determine the effects of progressive relaxation exercise and mindfulness meditation on dyspnea, fatigue and care dependency in patients with COPD. The present study investigates the effects of progressive muscle relaxation and mindfulness meditation in a single-site, 3-arm, assessor-blinded randomized, controlled study of 65 COPD patients. Arm 1: meditation; Arm 2: relaxation; Arm 3: Control.The investigators hypothesize that Progressive muscle relaxation and mindfulness meditation will decrease the severity of dyspnea, fatigue and care dependency.

ELIGIBILITY:
Inclusion Criteria:

* older than 40 years
* diagnosed with stage III-IV COPD
* had at least primary school degree
* had no cognitive dysfunction, or communication problems
* were residing in Ankara.

Exclusion Criteria:

* history of cognitive dysfunction, or communication problems
* illiteracy
* applying any complementary and integrative approach during the study
* participating in a pulmonary rehabilitation program during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in dyspnea | Baseline measurements, at the end of 12th week and four weeks after the completion of the interventions
  Dyspnea will be measured by The Dyspnea-12 Scale. The range of total score was from 0 to 36, with higher scores demonstrating higher dyspnea level.
Change in fatigue | Baseline measurements, at the end of 12th week and four weeks after the completion of the interventions
  Quality of live will be measured by Asthma Fatigue Scale (CAFS). The CAFS scores is standardized to 0-100 in line with the following formula, (100 × (total score-minimum value to be obtained)/range), with higher scores indicating greater fatigue.
Change in care dependency | Baseline measurements, at the end of 12th week and four weeks after the completion of the interventions
  Quality of live will be measured by Care Dependency Scale (CDS). The sum of the scores changes from 17 to 85, with higher scores demonstrating lower dependence.

OTHER OUTCOMES:
Dyspnea | Baseline
  The Dyspnea-12 Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided